CLINICAL TRIAL: NCT00254475
Title: A Study to Evaluate the Efficacy of the Valsartan/Simvastatin Combinations 160/20mg up Titrated to 320/20mg Versus 160/40mg up Titrated to 320/40mg in Patients With Both Essential Hypertension and Hypercholesterolemia
Brief Title: A Study to Evaluate the Efficacy of Valsartan/Simvastatin Combinations in Patients With Both Essential Hypertension and Hypercholesterolemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: CVAS489A2403
Record Dates: First submitted 2005-11-07; First posted 2005-11-16 (Estimated); Last update posted 2014-08-19 (Estimated); Status verified 2014-08

CONDITIONS: Essential Hypertension; Hypercholesterolemia
Keywords: Valsartan; simvastatin; hypertension; hypercholesterolemia; angiotensin II receptor blocker
MeSH Terms: conditions — Essential Hypertension; Hypercholesterolemia; Hypertension | interventions — Simvastatin; Valsartan

INTERVENTIONS:
Drug: simvastatin
Drug: valsartan

SUMMARY:
The purpose of this study is to provide data on the dose response of simvastatin in lowering LDL-C when it is co-administered with valsartan in patients with both essential hypertension and hypercholesterolemia. The primary objective of the study will be to show that the combination of valsartan 160mg/simvastatin 40mg has superior efficacy compared to the combination of valsartan 160mg/simvastatin 20mg in percentage change from baseline in LDL-C.

ELIGIBILITY:
Inclusion Criteria:

* Elevated LDL-Cholesterol
* Essential hypertension

Exclusion Criteria:

* Severe Hypertension
* Prior or known muscular or neuromuscular disease of any type
* A history of cardiovascular disease
* Hypertension or hypercholesterolemia due to secondary causes
* Uncontrolled diabetes or insulin treatment
* Evidence of hepatic or renal disease

Other protocol-defined exclusion criteria may apply

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 871 (Actual)
Dates: Start 2005-11; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Low density lipoproteins after 6 weeks

SECONDARY OUTCOMES:
Lipid profile at 6, 12 wks
BP < 140/90 mmHg in non diabetics, or < 130/80 mmHg in diabetics, and LDL-C < 2.6, 3.4 or 4.1 mmol/l based on risk group at 6, 12 wks
SBP < 140 mmHg in non diabetics, < 130 mmHg in diabetics, or 20 mmHg decrease in SBP from baseline and DBP < 90 mmHg in non diabetics, DBP < 80 mmHg in diabetics, or 10 mmHg decrease in DBP from baseline at 6, 12 wks
Systolic and diastolic bp at 6, 12 wks
Serious/adverse events, labs, physical exams, vitals up to 12 wks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceutical, Study Director — Novatis Pharmaceuticals
Locations (2):
- Investigative Centers, Germany
- Novartis Pharmaceuticals, Basel, Switzerland

REFERENCES:
- [Derived] Rump LC, Baranova E, Okopien B, Weisskopf M, Kandra A, Ferber P. Coadministration of valsartan 160 and 320 mg and simvastatin 20 and 40 mg in patients with hypertension and hypercholesterolemia: a multicenter, 12-week, double-blind, double-dummy, parallel-group superiority study. Clin Ther. 2008 Oct;30(10):1782-93. doi: 10.1016/j.clinthera.2008.10.004. PMID 19014834